CLINICAL TRIAL: NCT02900144
Title: Modified Comprehensive Behavioral Intervention for Tics: Treating Children With Tic Disorders, Co-occurring ADHD and Psychosocial Impairment
Brief Title: Modified Comprehensive Behavioral Intervention for Tics (M_CBIT)
Acronym: M_CBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erica Greenberg, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P001396
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Tourette Syndrome; ADHD
MeSH Terms: conditions — Tourette Syndrome; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified CBIT Treatment Arm (Experimental): In this arm, participants will receive the modified CBIT protocol. In addition to addressing tics, the treatment in this arm will also directly address ADHD symptoms using CBT for ADHD techniques, and quality of life concerns. The treatment itself will be modified to be more accessible to an ADHD population. The treatment will consist of twelve 50-min sessions: ten weekly and then two every other week for relapse prevention.
  Interventions: Behavioral: Modified Comprehensive Behavioral Intervention for Tics
- Standard CBIT Treatment Arm (Active Comparator): In this arm, participants will receive the standard CBIT intervention (Piacentini et al 2010). The primary components of CBIT are habit reversal training, relaxation training and a functional interventional to assess the environment for situations/factors that exacerbate or sustain tics. The treatment will consist of twelve 50-min sessions: ten weekly and then two every other week for relapse prevention.
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics

INTERVENTIONS:
Behavioral: Modified Comprehensive Behavioral Intervention for Tics — In this arm, participants will receive the modified CBIT protocol. In addition to addressing tics, the treatment in this arm will also directly address ADHD symptoms using CBT for ADHD techniques, and quality of life concerns. The treatment itself will be modified to be more accessible to an ADHD population. The treatment will consist of twelve 50-min sessions: ten weekly and then two every other week for relapse prevention.
  Arms: Modified CBIT Treatment Arm
Behavioral: Comprehensive Behavioral Intervention for Tics — In this arm, participants will receive the standard CBIT intervention (Piacentini et al 2010). The primary components of CBIT are habit reversal training, relaxation training and a functional interventional to assess the environment for situations/factors that exacerbate or sustain tics. The treatment will consist of twelve 50-min sessions: ten weekly and then two every other week for relapse prevention.
  Arms: Standard CBIT Treatment Arm

SUMMARY:
The main purpose of this trial is to develop and investigate the effects of a modified comprehensive behavioral intervention for tics (CBIT) protocol for children and adolescents with chronic tic disorders and ADHD.

CBIT is a first-line behavioral treatment for individuals with tic disorders. However, the benefit of CBIT is mitigated in those with co-occurring ADHD, as ADHD is negatively associated with effect size in behavioral treatments for tics. Additionally, while tic disorders are associated with reduced quality of life measures, CBIT is 'tic-specific.' Despite improving tics, measures do not show associated improved quality of life. Currently, there are no standardized behavioral treatments for tics that account for ADHD symptoms and/or addresses the impact that tics and ADHD symptoms have on quality of life.

The first aim is to develop a treatment protocol that combines elements from CBIT, Cognitive Behavioral Therapy (CBT) for ADHD and factors targeting psychosocial impairment.

The second aim is to determine the treatment feasibility and acceptability (e.g. retention, reasons for treatment refusal and dropout, and motivation) of this modified CBIT treatment. The investigators will evaluate and assess the randomization process, the treatment modules, and the expectations and satisfaction of the participants and their parents.

The final aim is to use a pilot randomized control trial (RCT) design to evaluate improvement using measures including tic, ADHD and quality of life scales as rated by a blinded clinician. Though the investigators will evaluate efficacy of the modified protocol, the primary purpose will remain feasibility. The hope is to use this study to develop larger trials in the future.

DETAILED DESCRIPTION:
Comprehensive behavior intervention for tics (CBIT) is a first-line behavioral treatment for individuals with tic disorders. However, the benefit of CBIT is mitigated in those with co-occurring ADHD, as ADHD is negatively associated with effect size in behavioral treatments for tics. Additionally, while tic disorders are associated with reduced quality of life measures, CBIT is 'tic-specific.' Despite improving tics, measures do not show associated improved quality of life. Currently, there are no standardized behavioral treatments for tics that account for ADHD symptoms and/or address the impact that tics and ADHD symptoms have on quality of life. The main purpose of this trial is to develop and then investigate the effects of a modified comprehensive behavioral intervention for tics (CBIT) protocol for children and adolescents with chronic tic disorders and ADHD.

Aim 1: Development a treatment protocol. The first aim is to develop a treatment protocol that combines elements from CBIT, Cognitive Behavioral Therapy (CBT) for ADHD, and factors targeting psychosocial impairment. A new treatment protocol, called "Living With Tics" was recently developed by Dr. Eric Storch et al to help improve quality of life in those with tic disorders. In addition to incorporating components of modules of the above listed treatments, the modules themselves will be adapted to be more accessible to those with ADHD. As tic disorders often have a significant impact on the family, the investigators will incorporate parent involvement into the treatment as well.

Aim 2: Treatment Feasibility and Acceptability. The investigators' second aim is to determine the treatment feasibility and acceptability of the developed protocol. They will examine the retention rates, reasons for treatment refusal and dropout, and subject/parents motivation for this modified CBIT treatment. They plan to evaluate and assess the randomization process, the treatment modules, and the expectations and satisfaction of the participants and their parents. They will use measures including expectancy and satisfaction scales, and Likert scales will be provided at the end of each session to help determine which components of the modules were most and/or least helpful. From those results, the investigators can continue to adapt the treatment protocol for future, larger studies.

Aim 3: Pilot test the treatment's effectiveness. The final aim is to conduct a pilot randomized control trial (RCT) to test the developed protocol in youth with tic disorders and co-morbid ADHD. Half the subjects will undergo treatment with the modified protocol, and half of the subjects will receive standard CBIT treatment. A broad range of outcome measures will be used to evaluate tic symptoms, ADHD symptoms, and quality of life, and predictors of treatment response will be explored. The following scales will be used: Yale Global Tic Severity Scale (YGTSS), NICHQ Vanderbilt Assessment Scales, and Pediatric Quality of Life Inventory-Child Version (PedsQL) scale, as rated by a blinded clinician. Additionally, the investigators will compare which components were most/least helpful to subjects. Though the investigators will evaluate efficacy of the modified protocol, the primary purpose will remain feasibility. The investigators hope to use this study to develop larger randomized controlled trials in the future.

The modified CBIT treatment will be based on the original CBIT protocol developed by Dr. John Piacentini et al in 2010, a CBT for ADHD in adolescents protocol recently developed by Dr. Susan Sprich et al, and Dr. Eric Storch's "Living with Tics" protocol. Techniques from other studies, which combined and adapted protocols will be incorporated as well.

The treatment will be divided into three phases: Evaluation/Psychoeducation, Basic Intervention, and Relapse Prevention, with a total of 12 sessions.

Prior to beginning the treatment, to make sure the subject qualifies, parent(s) and subject will be asked to come in to complete a baseline assessment component.

Evaluation/Psychoeducation (Sessions 1-2): The first 1-2 sessions will focus on assessing the subject's tics and ADHD symptoms, and assessing the impact of tics and ADHD on the subjects' lives. Psychoeducation about tics/Tourette Syndrome and ADHD, and the CBIT and CBT models will be provided. The therapist will create a hierarchy with the patient regarding which tics are most bothersome and what other symptoms/stressors are most impactful on everyday life. Planning and organizing skills and the idea of function-based interventions will also be introduced. Participants will be encouraged to bring their parent(s) to these initial assessment sessions to familiarize the parent(s) with the treatment methods and allow them to ask questions about tics and ADHD and/or the intervention. If appropriate, parents will be involved in the treatment or homework procedures, but this will vary depending on the comfort level and potential benefit as assessed for each child.

Basic Interventions (Session 3 to Session 10): Beginning in Session 3, basic CBIT, cognitive and behavioral methods will be taught during office sessions and assigned as homework throughout the treatment. In addition to including modules that will specifically target ADHD symptoms (such as those on organization and planning and distractibility), modules in general will be designed to target an ADHD population. Modules will include a combination of activity schedules, positive reinforcements to promote on-task behavior, short "brain breaks" in between activities, repetition of key concepts, and the use of visual aides during the sessions and between sessions at home. Handouts describing the topics covered will also be provided to the parent/patient at the conclusion of each session. Relaxation techniques will be incorporated. Some adapted modules from "Living with Tics" will be included depending on the patients' identified difficulties.

Relapse Prevention (Sessions 11-12): The final sessions, each spaced two weeks after the last session, will focus on relapse prevention. The purpose of the spaced sessions in to allow the patient to get more practice and learn to be their own therapist in between meetings. Residual problems and fears about ending treatment will be addressed, and unrealistically optimistic or pessimistic thoughts about treatment termination will be challenged. Patients will learn to anticipate possible symptom recurrence and its relationship to stress, mood, and other factors; counter negative thoughts about setbacks; and handle lapses and setbacks. Parents will also be encouraged to attend the last session(s) if the child/adolescent or clinician feels it would be appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Have a DSM-5-based diagnosis of Tourette Syndrome or Persistent Motor or Vocal Tic Disorder
2. Have a diagnosis of ADHD by DSM-5 standards, or a previous diagnosis of ADHD where there are some residual symptoms (at least 7/18) but does not currently meet diagnostic criteria due to current medications.
3. Tic disorder is the most problematic psychiatric disorder and the primary reason for seeking treatment
4. Have a current total tic severity score of >13 (or >9 if CTD) on the Yale Global Tic Severity Score (YGTSS), and a current total impairment score of >19 on the YGTSS
5. Be male or female and between 10-17 years of age at the start of the treatment, inclusive
6. Be able to communicate meaningfully with the investigators and be competent to provide written assent; both parental informed consent and adolescent assent must be obtained
7. Be English speaking

Exclusion Criteria:

1. Comorbid psychiatric diagnoses including: alcohol or substance abuse or dependence within the past 3 months, psychosis, organic mental disorder, current mania, developmental delay, estimated IQ <80 on the Wechsler Abbreviated Scale of Intelligence (WASI), other cognitive impairment that would interfere with ability to engage in CBT, or other developmental/cognitive impairment that precludes the participant from being able to communicate meaningfully with the treater
2. Those deemed to pose a serious suicidal or homicidal threat (e.g., suicide attempt within past 6 months and/or endorsement of "I want to kill myself" on the Children's Depression Inventory (CDI)).
3. Current illness (tics or otherwise) so severe that an immediate psychopharmacological evaluation is warranted
4. Any clinical features requiring a higher level of care than outpatient (as determined by evaluator).
5. Intent to travel for a period longer than two weeks (such that three sessions would be missed) during the proposed time-frame of the study. However, this criterion may be waived as per the discretion of the Principal investigator.
6. In general, the participant cannot be engaged in concurrent psychotherapy - if they are, they would need to stop (no lag time required between stopping current therapy and beginning this intervention). Decisions can be made on a case by case basis if the therapy is for a concern/disorder separate from mood, anxiety or OCD-spectrum disorders (e.g. gender dysphoria).
7. Four or more sessions of previous CBT treatment similar to the current treatment (CBIT and/or CBT for ADHD) within the last five years
8. Participants can be receiving psychotropic medication, but they must be on a stable dose for four weeks prior to the study baseline assessment and maintain this dosage throughout the course of the study. If a potential participant is taking psychotropic medication at the time of the phone evaluation or the first in-person study assessment and wishes to discontinue this medication to enter the trial, the participant will be asked to discuss this option with their prescribing physician to determine whether medication discontinuation would be safe and in the participant's best interest. We will not influence the decision or procedures participants choose with their prescribing physician. If the participant decides to discontinue treatment with the psychotropic medication, he/she must wait for four weeks before receiving a baseline assessment.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Questionnaire | 26 weeks
  Scale that measures the subject's satisfaction with the treatment
Expectancy Therapy Evaluation Form | Baseline
  Rates subject's expectations about effectiveness of the treatment
Satisfaction Scale for Module 1 | 1 week
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Expectancy Therapy Evaluation Form | 6 weeks
  Rates subject's expectations about effectiveness of the treatment
Satisfaction Scale for Module 2 | 2 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 3 | 3 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 4 | 4 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 5 | 5 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 6 | 6 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 7 | 7 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 8 | 8 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 9 | 9 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 10 | 10 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 11 | 12 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Satisfaction Scale for Module 12 | 14 weeks
  Brief Likert scale/multiple choice questions assessing the satisfaction/effectiveness of each session.
Patient Satisfaction Questionnaire | 6 weeks
  Scale that measures the patient's satisfaction with the treatment
Patient Satisfaction Questionnaire | 14 weeks
  Scale that measures the patient's satisfaction with the treatment

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale | Change from baseline to mid-point (6 weeks)
  Measures tic symptom severity and impairment
Yale Global Tic Severity Scale | Change from baseline to end-point (14 weeks)
  Measures tic symptom severity and impairment
Yale Global Tic Severity Scale | Change from baseline to 3months following end-point (26 weeks)
  Measures tic symptom severity and impairment
Vanderbilt Assessment Scale - ADHD | Change from baseline to mid-point (6 weeks)
  Measures DSM-IV ADHD and other externalizing behaviors
Vanderbilt Assessment Scale - ADHD | Change from baseline to end-point (14 weeks)
  Measures DSM-IV ADHD and other externalizing behaviors
Vanderbilt Assessment Scale - ADHD | Change from baseline to 3months following end-point (26 weeks)
  Measures DSM-IV ADHD and other externalizing behaviors
Clinical Global Impression - Improvement Scale | Change from baseline to one week
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to one week
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to two weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to two weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to three weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to three weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to four weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to four weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to five weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to five weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to six weeks (mid-point)
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to six weeks (mid-point)
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to seven weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to seven weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to eight weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to eight weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to nine weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to nine weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to ten weeks
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to ten weeks
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to twelve weeks (session 11)
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to twelve weeks (session 11)
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to fourteen weeks (session 12)
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to fourteen weeks (session 12)
  Measures severity of illness on a Likert scale
Clinical Global Impression - Improvement Scale | Change from baseline to 3months after end-point (26 weeks)
  Measures improvement on a Likert scale
Clinical Global Impression - Severity Scale | Change from baseline to 3months after end-point (26 weeks)
  Measures severity of illness on a Likert scale
Pediatric Quality of Life Inventory (PedsQL)-Child Version | Change from baseline to mid-point (6 weeks)
  Assesses pediatric population subject's quality of life on a scale of 0-100, with higher scores indicating a better quality of life.
Pediatric Quality of Life Inventory (PedsQL)-Child Version | Change from baseline to end-point (14 weeks)
  Assesses pediatric population subject's quality of life on a scale of 0-100, with higher scores indicating a better quality of life.
Pediatric Quality of Life Inventory (PedsQL)-Child Version | Change from baseline to 3months following end-point (26 weeks)
  Assesses pediatric population subject's quality of life on a scale of 0-100, with higher scores indicating a better quality of life.
Parent Tic Questionnaire (PTQ) | Mid-point (6 weeks)
  Measures severity of specific motor and vocal tics in terms of their frequency and intensity on a scale of 1-4, with higher scores indicating greater frequency and intensity.
Parent Tic Questionnaire (PTQ) | End-point (14 weeks)
  Measures severity of specific motor and vocal tics in terms of their frequency and intensity on a scale of 1-4, with higher scores indicating greater frequency and intensity.
Parent Tic Questionnaire (PTQ) | 3months following end-point (26 weeks)
  Measures severity of specific motor and vocal tics in terms of their frequency and intensity on a scale of 1-4, with higher scores indicating greater frequency and intensity.
ADHD - Self-report | Change from baseline to mid-point (6 weeks)
  Self-report of ADHD symptoms
ADHD - Self-report | Change from baseline to end-point (14 weeks)
  Self-report of ADHD symptoms
ADHD - Self-report | Change from baseline to 3months following end-point (26 weeks)
  Self-report of ADHD symptoms

OTHER OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale | Change from baseline to mid-point (6 weeks)
  Assesses severity of obsessive-compulsive symptoms in the last week
Children's Yale-Brown Obsessive Compulsive Scale | Change from baseline to end-point (14 weeks)
  Assesses severity of obsessive-compulsive symptoms in the last week
Children's Yale-Brown Obsessive Compulsive Scale | Change from baseline to 3months following end-point (26 weeks)
  Assesses severity of obsessive-compulsive symptoms in the last week
Children's Depression Inventory | Change from baseline to mid-point (6 weeks)
  Assesses depressive symptoms in children
Children's Depression Inventory | Change from baseline to end-point (14 weeks)
  Assesses depressive symptoms in children
Children's Depression Inventory | Change from baseline to 3months following end-point (26 weeks)
  Assesses depressive symptoms in children
Emotion Regulation Questionnaire | Change from baseline to mid-point (6 weeks)
  Measures emotion regulation strategies
Emotion Regulation Questionnaire | Change from baseline to end-point (14 weeks)
  Measures emotion regulation strategies
Emotion Regulation Questionnaire | Change from baseline to 3months following end-point (26 weeks)
  Measures emotion regulation strategies
Concomitant Medication and Therapy Questionnaire | 1 week
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 2 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 3 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 4 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 5 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 6 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 7 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 8 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 9 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 10 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 12 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
Concomitant Medication and Therapy Questionnaire | 14 weeks
  Tracks whether there are any concurrent therapy and/or medication changes
The Caregiver Strain Questionnaire | Change from baseline to mid-point (6 weeks)
  Assesses the extent to which the subject's condition has negatively affected the family
The Caregiver Strain Questionnaire | Change from baseline to end-point (14 weeks)
  Assesses the extent to which the subject's condition has negatively affected the family
The Caregiver Strain Questionnaire | Change from baseline to 3months following end-point (26 weeks)
  Assesses the extent to which the subject's condition has negatively affected the family
Child Tourette's Syndrome Impairment Scale | Change from baseline to mid-point (6 weeks)
  Assesses the impact that tics have on school, home, and social activities
Child Tourette's Syndrome Impairment Scale | Change from baseline to end-point (14 weeks)
  Assesses the impact that tics have on school, home, and social activities
Child Tourette's Syndrome Impairment Scale | Change from baseline to 3months following end-point (26 weeks)
  Assesses the impact that tics have on school, home, and social activities

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achenbach, T. M. (1991). Manual for the child behavior checklist/4-18 and 1991 Profile. Burlington: University of Vermont, Department of Psychiatry.
- [Background] Antshel KM, Faraone SV, Gordon M. Cognitive behavioral treatment outcomes in adolescent ADHD. J Atten Disord. 2014 Aug;18(6):483-95. doi: 10.1177/1087054712443155. Epub 2012 May 24. PMID 22628140
- [Background] "Attention Deficit Hyperactivity Disorder (ADHD)." Centers for Disease Control and Prevention - National Center for Health Statistics. 2015
- [Background] Barkley, R.A. (1990). Attention-deficit hyperactivity disorder: A handbook for diagnosis and treatment. New York, NY: Guilford Press.
- [Background] Borkovec TD, Nau SD: Credibility for analogue therapy rationales. J Behav Ther Exp Psychiatry 1972; 3:257-260
- [Background] Brannan AM, Heflinger CA, Bickman L. The Caregiver Strain Questionnaire: measuring the impact on the family of living with a child with serious emotional disturbance. J Emot Behav Disord. 1997;5(4):212-222
- [Background] Chang S, Himle M, Tucker B, Woods D, Piacentini J. Initial psychometric properties of a brief parent- report instrument for assessing tic severity in children with chronic tic disorders. Child Fam Behav Ther. 2009; 31(3):181-191.
- [Background] DuPaul, G.J., Power, T.J., Anastopoulos, A.D., & Reid, R. (1998). ADHD rating scale-IV: Checklists, norms, and clinical interpretations. New York, NY: Guilford Press
- [Background] Eddy CM, Cavanna AE, Gulisano M, Agodi A, Barchitta M, Cali P, Robertson MM, Rizzo R. Clinical correlates of quality of life in Tourette syndrome. Mov Disord. 2011 Mar;26(4):735-8. doi: 10.1002/mds.23434. Epub 2010 Nov 10. PMID 21506153
- [Background] El Malhany N, Gulisano M, Rizzo R, Curatolo P. Tourette syndrome and comorbid ADHD: causes and consequences. Eur J Pediatr. 2015 Mar;174(3):279-88. doi: 10.1007/s00431-014-2417-0. Epub 2014 Sep 17. PMID 25224657
- [Background] Fabiano GA, Pelham WE Jr, Coles EK, Gnagy EM, Chronis-Tuscano A, O'Connor BC. A meta-analysis of behavioral treatments for attention-deficit/hyperactivity disorder. Clin Psychol Rev. 2009 Mar;29(2):129-40. doi: 10.1016/j.cpr.2008.11.001. Epub 2008 Nov 11. PMID 19131150
- [Background] Guy W. ECDEU Assessment Manual for Psychopharmacology. Washington, DC, US Department of HEW Publications, 1976
- [Background] Halldorsdottir T, Ollendick TH, Ginsburg G, Sherrill J, Kendall PC, Walkup J, Sakolsky DJ, Piacentini J. Treatment Outcomes in Anxious Youth with and without Comorbid ADHD in the CAMS. J Clin Child Adolesc Psychol. 2015;44(6):985-91. doi: 10.1080/15374416.2014.952008. Epub 2014 Oct 13. PMID 25310142
- [Background] Hirschtritt ME, Lee PC, Pauls DL, Dion Y, Grados MA, Illmann C, King RA, Sandor P, McMahon WM, Lyon GJ, Cath DC, Kurlan R, Robertson MM, Osiecki L, Scharf JM, Mathews CA; Tourette Syndrome Association International Consortium for Genetics. Lifetime prevalence, age of risk, and genetic relationships of comorbid psychiatric disorders in Tourette syndrome. JAMA Psychiatry. 2015 Apr;72(4):325-33. doi: 10.1001/jamapsychiatry.2014.2650. PMID 25671412
- [Background] Jarrett MA, Ollendick TH. Treatment of comorbid attention-deficit/hyperactivity disorder and anxiety in children: a multiple baseline design analysis. J Consult Clin Psychol. 2012 Apr;80(2):239-44. doi: 10.1037/a0027123. Epub 2012 Feb 6. PMID 22309474
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Maric M, van Steensel FJA, Bogels SM. Parental Involvement in CBT for Anxiety-Disordered Youth Revisited: Family CBT Outperforms Child CBT in the Long Term for Children With Comorbid ADHD Symptoms. J Atten Disord. 2018 Mar;22(5):506-514. doi: 10.1177/1087054715573991. Epub 2015 Mar 9. PMID 25755259
- [Background] McGuire JF, Arnold E, Park JM, Nadeau JM, Lewin AB, Murphy TK, Storch EA. Living with tics: reduced impairment and improved quality of life for youth with chronic tic disorders. Psychiatry Res. 2015 Feb 28;225(3):571-9. doi: 10.1016/j.psychres.2014.11.045. Epub 2014 Dec 4. PMID 25500348
- [Background] McGuire JF, Nyirabahizi E, Kircanski K, Piacentini J, Peterson AL, Woods DW, Wilhelm S, Walkup JT, Scahill L. A cluster analysis of tic symptoms in children and adults with Tourette syndrome: clinical correlates and treatment outcome. Psychiatry Res. 2013 Dec 30;210(3):1198-204. doi: 10.1016/j.psychres.2013.09.021. Epub 2013 Sep 27. PMID 24144615
- [Background] McGuire JF, Piacentini J, Brennan EA, Lewin AB, Murphy TK, Small BJ, Storch EA. A meta-analysis of behavior therapy for Tourette Syndrome. J Psychiatr Res. 2014 Mar;50:106-12. doi: 10.1016/j.jpsychires.2013.12.009. Epub 2013 Dec 28. PMID 24398255
- [Background] McGuire JF, Ricketts EJ, Piacentini J, Murphy TK, Storch EA, Lewin AB. Behavior Therapy for Tic Disorders: An Evidenced-based Review and New Directions for Treatment Research. Curr Dev Disord Rep. 2015 Dec;2(4):309-317. doi: 10.1007/s40474-015-0063-5. Epub 2015 Sep 14. PMID 26543797
- [Background] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Background] Rapee, R. M., Wignall, A., Hudson, J. L., & Schniering, C. A. (2000). Treating anxious children and adolescents: An evidence-based approach. Oakland, CA: New Harbringer
- [Background] Ricketts EJ, Gilbert DL, Zinner SH, Mink JW, Lipps TD, Wiegand GA, Vierhile AE, Ely LJ, Piacentini J, Walkup JT, Woods DW. Pilot Testing Behavior Therapy for Chronic Tic Disorders in Neurology and Developmental Pediatrics Clinics. J Child Neurol. 2016 Mar;31(4):444-50. doi: 10.1177/0883073815599257. Epub 2015 Aug 13. PMID 26271790
- [Background] Rowe J, Yuen HK, Dure LS. Comprehensive behavioral intervention to improve occupational performance in children with Tourette disorder. Am J Occup Ther. 2013 Mar-Apr;67(2):194-200. doi: 10.5014/ajot.2013.007062. PMID 23433274
- [Background] Safren SA, Otto MW, Sprich S, Winett CL, Wilens TE, Biederman J. Cognitive-behavioral therapy for ADHD in medication-treated adults with continued symptoms. Behav Res Ther. 2005 Jul;43(7):831-42. doi: 10.1016/j.brat.2004.07.001. PMID 15896281
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of diagnosed Tourette syndrome in persons aged 6-17 years - United States, 2007. MMWR Morb Mortal Wkly Rep. 2009 Jun 5;58(21):581-5. PMID 19498335
- [Background] Scahill L, Riddle MA, McSwiggin-Hardin M, Ort SI, King RA, Goodman WK, Cicchetti D, Leckman JF. Children's Yale-Brown Obsessive Compulsive Scale: reliability and validity. J Am Acad Child Adolesc Psychiatry. 1997 Jun;36(6):844-52. doi: 10.1097/00004583-199706000-00023. PMID 9183141
- [Background] Scahill L, Specht M, Page C. The Prevalence of Tic Disorders and Clinical Characteristics in Children. J Obsessive Compuls Relat Disord. 2014 Oct 1;3(4):394-400. doi: 10.1016/j.jocrd.2014.06.002. PMID 25436183
- [Background] Scahill L, Woods DW, Himle MB, Peterson AL, Wilhelm S, Piacentini JC, McNaught K, Walkup JT, Mink JW. Current controversies on the role of behavior therapy in Tourette syndrome. Mov Disord. 2013 Aug;28(9):1179-83. doi: 10.1002/mds.25488. Epub 2013 May 16. PMID 23681719
- [Background] Scharf JM, Miller LL, Gauvin CA, Alabiso J, Mathews CA, Ben-Shlomo Y. Population prevalence of Tourette syndrome: a systematic review and meta-analysis. Mov Disord. 2015 Feb;30(2):221-8. doi: 10.1002/mds.26089. Epub 2014 Dec 8. PMID 25487709
- [Background] Sciberras E, Mulraney M, Anderson V, Rapee RM, Nicholson JM, Efron D, Lee K, Markopoulos Z, Hiscock H. Managing Anxiety in Children With ADHD Using Cognitive-Behavioral Therapy: A Pilot Randomized Controlled Trial. J Atten Disord. 2018 Mar;22(5):515-520. doi: 10.1177/1087054715584054. Epub 2015 May 4. PMID 25939582
- [Background] Sheehan DV, Sheehan KH, Shytle RD, Janavs J, Bannon Y, Rogers JE, Milo KM, Stock SL, Wilkinson B. Reliability and validity of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). J Clin Psychiatry. 2010 Mar;71(3):313-26. doi: 10.4088/JCP.09m05305whi. PMID 20331933
- [Background] Silverman WK, Saavedra LM, Pina AA. Test-retest reliability of anxiety symptoms and diagnoses with the Anxiety Disorders Interview Schedule for DSM-IV: child and parent versions. J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):937-44. doi: 10.1097/00004583-200108000-00016. PMID 11501694
- [Background] Specht MW, Woods DW, Piacentini J, Scahill L, Wilhelm S, Peterson AL, Chang S, Kepley H, Deckersbach T, Flessner C, Buzzella BA, McGuire JF, Levi-Pearl S, Walkup JT. Clinical Characteristics of Children and Adolescents with a Primary Tic Disorder. J Dev Phys Disabil. 2011 Feb;23(1):15-31. doi: 10.1007/s10882-010-9223-z. PMID 24999300
- [Background] Sprich SE, Knouse LE, Cooper-Vince C, Burbridge J, Safren SA. Description and Demonstration of CBT for ADHD in Adults. Cogn Behav Pract. 2012 Feb 1;17(1):10.1016/j.cbpra.2009.09.002. doi: 10.1016/j.cbpra.2009.09.002. PMID 24379644
- [Background] Sprich SE, Safren SA, Finkelstein D, Remmert JE, Hammerness P. A randomized controlled trial of cognitive behavioral therapy for ADHD in medication-treated adolescents. J Child Psychol Psychiatry. 2016 Nov;57(11):1218-1226. doi: 10.1111/jcpp.12549. Epub 2016 Mar 17. PMID 26990084
- [Background] Storch EA, Lack CW, Simons LE, Goodman WK, Murphy TK, Geffken GR. A measure of functional impairment in youth with Tourette's syndrome. J Pediatr Psychol. 2007 Sep;32(8):950-9. doi: 10.1093/jpepsy/jsm034. Epub 2007 May 23. PMID 17522110
- [Background] Storch EA, Merlo LJ, Lack C, Milsom VA, Geffken GR, Goodman WK, Murphy TK. Quality of life in youth with Tourette's syndrome and chronic tic disorder. J Clin Child Adolesc Psychol. 2007 Apr-Jun;36(2):217-27. doi: 10.1080/15374410701279545. PMID 17484694
- [Background] Storch EA, Morgan JE, Caporino NE, Brauer L, Lewin AB, Piacentini J. Psychosocial Treatment to Improve Resilience and Reduce Impairment in Youth With Tics: An Intervention Case Series of Eight Youth. Journal of Cognitive Psychotherapy 2012; 26(1):57-70
- [Background] U.S. Census Bureau
- [Background] Varni JW, Burwinkle TM, Seid M, Skarr D. The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr. 2003 Nov-Dec;3(6):329-41. doi: 10.1367/1539-4409(2003)0032.0.co;2. PMID 14616041
- [Background] Woods DW, Piacentini J, Himle MB, Chang S. Premonitory Urge for Tics Scale (PUTS): initial psychometric results and examination of the premonitory urge phenomenon in youths with Tic disorders. J Dev Behav Pediatr. 2005 Dec;26(6):397-403. doi: 10.1097/00004703-200512000-00001. PMID 16344654
- [Background] Woods DW, Piacentini JC, Scahill L, Peterson AL, Wilhelm S, Chang S, Deckersbach T, McGuire J, Specht M, Conelea CA, Rozenman M, Dzuria J, Liu H, Levi-Pearl S, Walkup JT. Behavior therapy for tics in children: acute and long-term effects on psychiatric and psychosocial functioning. J Child Neurol. 2011 Jul;26(7):858-65. doi: 10.1177/0883073810397046. Epub 2011 May 9. PMID 21555779
- [Background] Zhu Y, Leung KM, Liu PZ, Zhou M, Su LY. Comorbid behavioural problems in Tourette's syndrome are positively correlated with the severity of tic symptoms. Aust N Z J Psychiatry. 2006 Jan;40(1):67-73. doi: 10.1080/j.1440-1614.2006.01745.x. PMID 16403042
- [Background] Gullone E, Taffe J. The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): a psychometric evaluation. Psychol Assess. 2012 Jun;24(2):409-17. doi: 10.1037/a0025777. Epub 2011 Oct 24. PMID 22023559
- [Background] Kovacs M. Children's Depression Inventory (CDI). Toronto, Ontario, Canada: Multi-Health System. Inc; 1992.
- [Background] Rosler M, Retz W, Retz-Junginger P, Thome J, Supprian T, Nissen T, Stieglitz RD, Blocher D, Hengesch G, Trott GE. [Tools for the diagnosis of attention-deficit/hyperactivity disorder in adults. Self-rating behaviour questionnaire and diagnostic checklist]. Nervenarzt. 2004 Sep;75(9):888-95. doi: 10.1007/s00115-003-1622-2. German. PMID 15378249
- [Background] Steinberg EA, Drabick DA. A Developmental Psychopathology Perspective on ADHD and Comorbid Conditions: The Role of Emotion Regulation. Child Psychiatry Hum Dev. 2015 Dec;46(6):951-66. doi: 10.1007/s10578-015-0534-2. PMID 25662998
- [Background] Vanderbilt Assessment Scale. American Academy of Pediatrics and National Initiative for Children's Healthcare Quality. McNeil, 2002
- [Background] Wechsler D. (1999). Wechsler Abbreviated Scale of Intelligence (WASI). San Antonio, TX: Psychological Corporation.
- [Background] World Health Organization. Childhood ADHD Symptoms Scale Self-Report.